CLINICAL TRIAL: NCT01798875
Title: Effects of Different Therapies on Surrogate Markers of Cardiovascular Risk in Women With Polycystic Ovary Syndrome (PCOS)
Brief Title: PCOS, Therapy and Markers of Cardiovascular Risk
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Medical University of Gdansk (Other)
Responsible Party: Principal Investigator, Dominik Rachon, M.D. PhD, Medical University of Gdansk
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: POLovaRIS
Record Dates: First submitted 2013-02-22; First posted 2013-02-26 (Estimated); Last update posted 2013-03-01 (Estimated); Status verified 2013-02

CONDITIONS: PCOS
Keywords: pcos; metformin; oral contraception; cyproterone acetate
MeSH Terms: conditions — Polycystic Ovary Syndrome | interventions — Metformin; Contraceptives, Oral

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Metformin (Active Comparator): oral metformin at a dose of 850mg twice daily
  Interventions: Drug: oral metformin
- Oral contraceptive (Active Comparator): oral contraceptive containing 35ug of ethynylestradiol and 2mg of cyproterone acetate (21 day regimen)
  Interventions: Drug: oral contraceptive

INTERVENTIONS:
Drug: oral metformin
  Arms: Metformin
Drug: oral contraceptive
  Arms: Oral contraceptive

SUMMARY:
In addition to chronic anovulation and hyperandrogenemia, polycystic ovary syndrome (PCOS) is also characterized by peripheral insulin resistance and hyperinsulinaemia, which in turn lead to the development of diabetes, hypertension, atherosclerosis and coronary heart disease. Serum markers of inflammation are being increasingly recognized as predictors of atherosclerosis and cardiovascular risk, and chronic low-grade inflammation has been recently proposed to play a role in the pathogenesis of metabolic syndrome and type 2 diabetes mellitus. Therefore, the aim of the present study is to evaluate the effects of commonly used non-pharmacologic (diet and lifestyle change) and pharmacologic (oral contraceptives, metformin, anti-androgens) treatment strategies on classical and surrogate cardiovascular risk markers in women with PCOS. The study hypothesis is that some of the commonly used therapies of women with PCOS may have more favorable effects on classical and surrogate markers of cardiovascular risk then others or some of them may even confer a higher risk of cardiovascular events

ELIGIBILITY:
Inclusion Criteria:

* PCOS

Exclusion Criteria:

* diabetes
* pregnancy
* contraindications to oral contraceptives

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Estimated)
Dates: Start 2012-04; Primary Completion 2015-12 (Estimated); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
serum C-reactive protein (CRP) levels | 6 months

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Clinical and Experimental Endocrinology, Medical University of Gdansk, Gdansk, Poland

REFERENCES:
- [Derived] Dardzinska JA, Rachon D, Kuligowska-Jakubowska M, Aleksandrowicz-Wrona E, Ploszynski A, Wyrzykowski B, Lysiak-Szydlowska W. Effects of metformin or an oral contraceptive containing cyproterone acetate on serum c-reactive protein, interleukin-6 and soluble vascular cell adhesion molecule-1 concentrations in women with polycystic ovary syndrome. Exp Clin Endocrinol Diabetes. 2014 Feb;122(2):118-25. doi: 10.1055/s-0033-1363261. Epub 2014 Feb 19. PMID 24554512